CLINICAL TRIAL: NCT01562483
Title: The Analgesic Efficacy of Δ9-THC (Namisol®) in Patients With Persistent Postsurgical Abdominal Pain; a Randomized, Double Blinded, Placebo-controlled, Experiment
Brief Title: The Analgesic Efficacy of Δ9-THC (Namisol®) in Patients With Persistent Postsurgical Abdominal Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HEEL-2011-03
Record Dates: First submitted 2012-03-07; First posted 2012-03-23 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Postsurgical Pain; Abdominal Pain; Chronic Pain
Keywords: postsurgical pain; abdominal pain; visceral pain; chronic pain
MeSH Terms: conditions — Pain, Postoperative; Abdominal Pain; Chronic Pain; Visceral Pain | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- delta-9-tetrahydrocannabinol (namisol) (Experimental)
  Interventions: Drug: Tetrahydrocannabinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetrahydrocannabinol — The add-on treatment consists of two phases: a step-up phase (day 1-5: 3 mg TID; day 6-10: 5 mg TID), and a stable dose phase (day 11-52: 8 mg TID). The dosage may be tapered to at least 5 mg TID, when 8 mg is not tolerated.
  Other Names: Namisol; Dronabinol
  Arms: delta-9-tetrahydrocannabinol (namisol)
Drug: Placebo — Identical to the Namisol arm.
  Arms: Placebo

SUMMARY:
Persistent postsurgical abdominal pain (PPAP) is a very difficult to treat pain. This pain can persist for months or even years and significantly diminishes quality of life. The exact underlying cause for this pain persistence is still unclear, which makes its treatment still a challenge. The promising analgesic effects of Δ9-THC in previous research, plus the improved bioavailability of Namisol® in comparison with previous Δ9-THC substances form the basis of the present research proposal.

The current study aims to investigate the analgesic efficacy of Namisol® as add-on analgesic during a long-term treatment (52 days) of persistent postsurgical abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Pain should have developed after a surgical procedure
* Pain duration exceeding 3 months, and average NRS≥3
* Stable doses intake of analgesics for the past 2 months
* The patient has been informed about the study, understood the information and signed the informed consent form

Exclusion Criteria:

* Diagnosed irritated bowel syndrome (IBS) or chronic pancreatitis
* Patient took cannabinoids on a regular basis for at least one year
* Patient does not feel a pinprick test in the lower extremities
* Patient has a body mass index (BMI) above 36,0 kg/m2
* Patient suffers from serious painful conditions other than chronic pancreatitis
* Patient has a significant medical disorder that may interfere with the study or may pose a risk for the patient
* Patient uses any kind of concomitant medication that may interfere with the study or may pose a risk for the patient
* Patient does not tolerate oral intake of medication or liquids, or is refrained from oral intake because of medical reasons
* Patient demonstrates clinical relevant deviations in the electrocardiogram (ECG)
* Patient has an actual moderate to severe renal impairment
* Patient has an actual moderate to severe hepatic impairment
* Patient has a presence or history of major psychiatric illness
* Patient has experienced an epileptic seizure in the past
* Patient demonstrates clinically significant laboratory abnormalities
* Patient demonstrates a positive urine drug screen for THC, cocaine, MDMA, and amphetamines
* Patient demonstrates a positive test result on hepatitis B surface antigen, hepatitis C antibody or HIV antibody test
* Patient has a history of sensitivity / idiosyncrasy to THC
* Patient has a known or suspected lactose intolerance
* Female patient is pregnant or breastfeeding
* Patient intends to conceive a child during the course of the study
* Patient participates in another investigational drug study
* Patient has a clinical significant exacerbation in illness
* Patient is unwilling or unable to comply with the lifestyle guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Average VAS pain | Baseline versus day 52
  The primary outcome measure is defined as the reduction in average VAS pain scores at the end of the study (day 50-52) compared to the pre-treatment level between the Namisol® and placebo group, measured by a Visual Analoge Scale (VAS) in a pain diary.

SECONDARY OUTCOMES:
Electroencephalogram (EEG) | Baseline versus day 52
  Evoked potentials to noxious electrical stimuli, evoked potentials to auditory stimuli (oddball), and spontaneous brain activity will be measured in the electroencephalogram (EEG).
Quantitative Sensory Testing (QST) | Baseline versus day 15 and day 52
  Pressure pain thresholds, electrical thresholds, electric wind-up response, and Diffuse Noxious Inhibitory Control (DNIC) will be measured using Quantitative Sensory Testing (QST).
Depression and (pain related) anxiety | Baseline versus day 52
  Depression and (pain related) anxiety measured by questionnaires.
Pharmacodynamic parameters | Baseline versus day 15 and day 52
  Pharmacodynamics measured by body sway and questionnaires (VASBond & Lader and VASBowdle)
Safety parameters | Baseline until follow-up (day 59-61)
  * Laboratory
  * Electrocardiogram (ECG)
  * Heart Frequency (HF) / Blood Pressure (BP)
  * Adverse Events (AE)
Quality of life | Baseline versus day 52
  Quality of life will be evaluated by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, department of surgery
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] de Vries M, van Rijckevorsel DCM, Vissers KCP, Wilder-Smith OHG, van Goor H; Pain and Nociception Neuroscience Research Group. Tetrahydrocannabinol Does Not Reduce Pain in Patients With Chronic Abdominal Pain in a Phase 2 Placebo-controlled Study. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1079-1086.e4. doi: 10.1016/j.cgh.2016.09.147. Epub 2016 Oct 5. PMID 27720917